CLINICAL TRIAL: NCT05493579
Title: "Impact of Mandibular Implant Supported Overdenture on Changes of Electromyographic Activity, Brain Activity, Cognitive Function, Nutrition and Depression Status."
Brief Title: Impact of Implant Supported Overdenture on Changes of Electromyographic and Brain Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Noha Taha Kamel Taha Alloush, Assistant Lecturer, Misr International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC-PR-21-08
Record Dates: First submitted 2022-01-09; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-01

CONDITIONS: Implant Supported Overdenture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complete denture then complete implant supported overdenture (Experimental)
  Interventions: Other: Implant supported overdenture

INTERVENTIONS:
Other: Implant supported overdenture — Implant supported overdenture compared to complete denture

SUMMARY:
The purpose of this study is to evaluate and compare the effects of a mandibular implant-supported overdenture with a mandibular complete denture on electromyographic activity, brain activity, and cognitive performance in edentulous patients. Ten patients who are entirely edentulous and did not wear dentures will be chosen. To assess brain activity and cognitive function, electroencephalograms, the Mini-Mental State Examination (MMSE), and electromyographic examinations of the temporalis and masseter muscles will be performed prior to complete denture construction, one and three months after complete denture construction, and one and three months after implant supported overdenture insertion, respectively.

ELIGIBILITY:
Inclusion Criteria:

* All patients' ridges should be covered with firm mucosa which is free from any signs of inflammation or ulceration.
* Patients should be free from any bone disorder and exhibit adequate height and width of the residual alveolar ridge.
* All patients must have sufficient inter arch space.

Exclusion Criteria:

* Patients with oral or systemic diseases.
* Patients with xerostomia or excessive salivation.
* Patients with parafunctional habits (bruxism or clenching).
* Heavy smoker or alcoholic patients.
* Patients with history of temporo-mandibular dysfunction.
* Patients with neurological or psychiatric disorders.

Ages: 65 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Brain Activity (EEG) | 3 months
  An assessment of the patient's brain activity will be done. The waves obtained during all phases of assessment will be analyzed, and the software will separate the alpha waves, which occur in the frequency range of 8-12 Hz, evaluating their amplitude. The mean amplitude (in microvolts) of alpha waves was obtained.

SECONDARY OUTCOMES:
Cognitive Function (MMSE) | 3 months
  Cognitive function will be assessed using the Mini-Mental State Examination (MMSE) questionnaire. The MMSE set, with a total score of 30, assesses different domains of cognitive function. The MMSE comprises 30 questions, with 10 devoted to orientation; three items requiring registration of new information; five questions addressing attention and calculation; three recall items; eight items assessing language skills; and one construction question. Any score of 24 or more (out of 30) indicates normal cognition. Scores below this indicate severe (9 points), moderate (10-18 points), or mild (19-23 points) cognitive impairment.

OTHER OUTCOMES:
Muscle Activity (EMG) | 3 months
  The highest EMG activity in the masseter muscle and the anterior temporalis muscle will be calculated during the maximum clenching, maximal voluntary contraction (MVC) in the intercuspal position. The EMG signals will be stored and analyzed as root mean square (RMS) values expressed in microvolts (μV) and the mean amplitude of the motor unit potential (MUP) will be calculated in microvolts (μV).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry. AL Azhar University for Girls, Cairo, Egypt., Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided